CLINICAL TRIAL: NCT05412030
Title: A Phase 2, Randomized, Double-blind, Multi-dose, Dose Finding Study to Evaluate the Safety, Tolerability and Immunogenicity of AFX3772 Compared With PCVs in Healthy Infants
Brief Title: A Phase 2 Study to Evaluate the Safety, Tolerability, and Immune Response of AFX3772 Vaccine in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 219651; 2023-000423-36 (EudraCT Number)
Record Dates: First submitted 2022-06-03; First posted 2022-06-09 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Pneumonia, Bacterial; Pneumococcal Infections; Pneumonia, Pneumococcal
Keywords: Pneumonia, Pneumococcal; Infections; Streptococcal Infections; Pneumonia
MeSH Terms: conditions — Pneumonia, Bacterial; Pneumococcal Infections; Pneumonia, Pneumococcal; Infections; Streptococcal Infections; Pneumonia | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 Group 1 (Experimental): Infants are scheduled to receive up to three doses of 1 mcg AFX3772 as part of the primary series, followed by a booster dose. Those who do not receive the planned AFX3772 dose are administered PCV13 as standard of care (SOC).
  Interventions: Biological: AFX3772; Biological: Prevnar 13
- Part 1 Group 2 (Experimental): Infants are scheduled to receive up to three doses of 2 mcg AFX3772 as part of the primary series, followed by a booster dose. Those who do not receive the planned AFX3772 dose are administered PCV13 as SOC.
  Interventions: Biological: AFX3772; Biological: Prevnar 13
- Part 1 Group 3 (Experimental): Infants are scheduled to receive up to three doses of 5 mcg AFX3772 as part of the primary series, followed by a booster dose. Those who do not receive the planned AFX3772 dose are administered PCV13 as SOC.
  Interventions: Biological: AFX3772; Biological: Prevnar 13
- Part 1 Group 4 (Active Comparator): PCV13 administered intramuscularly within 12 months.
  Interventions: Biological: Prevnar 13
- Part 2 Group 5 (Experimental): Infants are scheduled to receive up to three doses of 2 mcg AFX3772 as part of the primary series, followed by a booster dose. Those who do not receive the planned AFX3772 dose are administered PCV20 as SOC.
  Interventions: Biological: AFX3772; Biological: Prevnar 20
- Part 2 Group 6 (Experimental): Infants are scheduled to receive up to three doses of 5 mcg AFX3772 as part of the primary series, followed by a booster dose. Those who do not receive the planned AFX3772 dose are administered PCV20 as SOC.
  Interventions: Biological: AFX3772; Biological: Prevnar 20
- Part 2 Group 7 (Active Comparator): PCV20 administered intramuscularly within 12 months.
  Interventions: Biological: Prevnar 20

INTERVENTIONS:
Biological: AFX3772 — AFX3772 administered intramuscularly.
  Arms: Part 1 Group 1; Part 1 Group 2; Part 1 Group 3; Part 2 Group 5; Part 2 Group 6
Biological: Prevnar 13 — PCV13 administered intramuscularly.
  Other Names: PCV13
  Arms: Part 1 Group 1; Part 1 Group 2; Part 1 Group 3; Part 1 Group 4
Biological: Prevnar 20 — PCV 20 administered intramuscularly.
  Other Names: PCV20
  Arms: Part 2 Group 5; Part 2 Group 6; Part 2 Group 7

SUMMARY:
This is a Phase 2 clinical study to support the use of AFX3772 in healthy infants for the prevention of pneumococcal disease. The purpose of this study is to determine the safety, tolerability, and immunogenicity of 3 different formulations of AFX3772 compared with Prevnar 13 (PCV13) and Prevnar 20 (PCV).

Part 1 is the dose escalation, lead-in portion of the study in which infants at each dose level will be randomized 3:1 in sequential cohorts of increasing doses of AFX3772 or PCV13.

In Part 2, infants will be randomized to receive either one of two dose levels of AFX3772 or PCV20.

ELIGIBILITY:
Inclusion Criteria:

• Is a full-term infant approximately 2 months of age at time of obtaining the informed consent.

Exclusion Criteria:

* Had prior administration of any pneumococcal vaccine.
* Has a known or suspected hypersensitivity to AFX3772, PCV13, PCV20 or any components of the formulations used.
* Has a known or suspected immunodeficiency or other conditions associated with immunosuppression that may require immunosuppressive drugs. In addition, the participant's biological mother has known HIV infection or known to be hepatitis B surface antigen positive.
* Has any clinically significant allergic condition or history prior to the first vaccination for primary immunization series.
* Has a history of microbiologically proven invasive disease caused by S. pneumoniae.
* Has received immunoglobulins.
* Has a bleeding diathesis or condition associated with prolonged bleeding that would contraindicate intramuscular injection.
* Has received systemic corticosteroids for a period of more than 14 days and has not completed the treatment for at least 30 days before study vaccine.

Ages: 42 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 388 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with solicited injection site events | Day 1 through Day 7 post-vaccination
  The assessed solicited injection site events are tenderness, redness/erythema and swelling.
Percentage of participants with solicited systemic events | Day 1 through Day 7 post-vaccination
  The assessed solicited systemic events are irritability, fever, decrease of appetite, increased sleep, and decrease in sleep.
Percentage of participants with AEs | Day 1 through Day 30
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention.
Percentage of participants with serious adverse events (SAEs) | Day 1 through 6 months post dose three
  An SAE is any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires in patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity.
  Medical or scientific judgment will be exercised by the investigator in deciding whether SAE reporting is appropriate in other situations such as significant medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition.

SECONDARY OUTCOMES:
Percentage of participants with a pneumococcal serotype-specific Immunoglobulin G (IgG) concentration of greater than or equal to (>=) 0.35 μg/mL or corresponding threshold | 30 days post-dose two, 30 days post-dose three
  Immunological responses were assessed in terms of percentage of participants with a pneumococcal serotype-specific IgG concentration >= 0.35 μg/mL or corresponding threshold.
Geometric mean concentration for serotype-specific IgG | 30 days post-dose two, 30 days post-dose three
  Immunological responses were assessed in terms of IgG GMCs and expressed as titers.

CONTACTS AND LOCATIONS:
Locations (42):
- United States (38):
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Saint Augustine, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Haughton, Louisiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Mankato, Minnesota
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Hastings, Nebraska
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Cranberry Township, Pennsylvania
  - GSK Investigational Site, Jefferson Hills, Pennsylvania
  - GSK Investigational Site, N. Huntingdon, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Brownsville, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Dickinson, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, McAllen, Texas
  - GSK Investigational Site, Richmond, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, Syracuse, Utah
  - GSK Investigational Site, Norfolk, Virginia
- Puerto Rico (4):
  - GSK Investigational Site, Bayamón
  - GSK Investigational Site, Caguas
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, San Juan

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf